CLINICAL TRIAL: NCT05476666
Title: Peripheral Venous Pressure as an Indicator of Central Venous Pressure in Post Operative Surgical Patients: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Navy Station Shifa Hospital (Other)
Responsible Party: Principal Investigator, Kenan Anwar Khan, Graded Anaesthetist, Principal Investigator, Pakistan Navy Station Shifa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ERC/2022/ANS/1
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Peripherial Venous Pressure; Central Venous Pressure; Fluid/Volume Status Monitoring of Patient
Keywords: Peripherial venous pressure; Central venous pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pressures measured (Experimental): Venous pressure measured through a peripherial and a central venous catheter/cannula
  Interventions: Procedure: Peripherial and central venous access

INTERVENTIONS:
Procedure: Peripherial and central venous access — Passing a peripherial and a central venous catheter/cannula

SUMMARY:
The study is aimed at comparing peripherial venous pressure as an indicator of central venous pressure in post operative surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA I/II/III surgical patients who require central venous access as part of their surgical treatment plan with no organ support in post operative period.
* Age between 18 and 75 years
* Who have atleast 1 x 18 gauge peripherial venous cannula in the upper limb from elbow below to the hand
* Who have given consent

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Peripherial venous pressure as an indicator of central venous pressure | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenan Khan, Principal Investigator — Pakistan Navy Station Shifa Hospital
Locations (1):
- PNS Shifa Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No